CLINICAL TRIAL: NCT06882122
Title: Neurophysiological and Biomolecular Effects of Atogepant in High Frequency Episodic Migraine (ATOM Project)
Brief Title: Neurophysiological and Biomolecular Effects of Atogepant in Episodic Migraine
Acronym: ATOM
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ATOM
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Migraine Disorder; Episodic Migraine
Keywords: Migraine; Gepants; endocannabinoid system; MicroRNAs; Habituation deficit; Central sensitization; Functional Connectivity
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HFEM group: High-frequency episodic migraine patients (8-14 migraine days per months) undergoing atogepant 60 mg daily for 3 months
  Interventions: Drug: Atogepant 60 mg

INTERVENTIONS:
Drug: Atogepant 60 mg — Atogepant 60 mg daily for 3 months

SUMMARY:
The investigators aim to assess and compare neurophysiological and biochemical changes induced by a 3-month treatment with atogepant (60 mg daily) in patients with high-frequency episodic migraine (8-14 monthly migraine days). Evaluations will include neurophysiological assessments (High-Density EEG, nociceptive reflexes, and visual evoked potentials) and biomolecular profiling (gene expression of endocannabinoid catabolizing enzymes, CGRP and PACAP plasma levels, and headache-specific microRNAs). Outputs will contribute to defining predictors of atogepant response, elucidating its effects on brain connectivity, excitability, and CGRP/endocannabinoid pathways, and identifying alternative therapeutic targets for non-responders.

DETAILED DESCRIPTION:
BACKGROUND:

Migraine is a highly prevalent neurological disease associated to a severe burden for patients and society. Despite recent advances, the knowledge of the molecular and biochemical pathways that turn on and off a migraine attack and lead to an increased frequency of attacks is still limited. In addition, the lack of predictors of the therapeutic response is a barrier to access to care and to a personalized approach. In recent years, several migraine-specific drugs have become available for the preventive treatment of the disease, which is aimed at reducing the frequency and the intensity of the attacks. Among the drugs currently available for migraine treatment, there are molecules that directly interfere with the calcitonin gene-related peptide (CGRP) pathway. Gepants, oral drugs that are CGRP receptor antagonists, represent a recently available pharmacological class for the acute and preventive treatment of migraines due to their specific mechanism of action.

The potential mechanism underlying the therapeutic benefit derived from drugs that block CGRP, as well as their impact on various biochemical and functional parameters associated with migraine pathophysiology, remains a topic of debate.

The objective of the ATOM project is to characterize the neurophysiological and biomolecular mechanisms underlying the therapeutic action of Atogepant (ATO), a drug belonging to the new pharmacological class of gepants. ATO has been shown to be effective in the preventive treatment of both chronic and episodic migraine. However, preventive treatment with gepants is still ineffective (reducing the number of monthly migraine days by less than 50%) in 30% of patients. This finding suggests that other biological pathways independent of CGRP may play a role in migraine pathophysiology. Among these, the endocannabinoid system has gained increasing importance over the years.

From a neurofunctional perspective, central sensitization is a significant aspect of migraine pathophysiology. Our group has demonstrated the utility of the nociceptive withdrawal reflex at the lower limb (RIII) in studying central sensitization. A subsequent study showed improvement in RIII reflex parameters in 30% of chronic migraine patients who responded to Erenumab after three months of treatment, suggesting a potential correlation between improved central sensitization and clinical benefit from anti-CGRP antibody treatment.

Additionally, migraine patients exhibit altered responses following repeated cranial stimulation, specifically a deficit in habituation to such stimuli. It has been described that the habituation pattern follows a characteristic course throughout the migraine cycle. The habituation deficit has been demonstrated through various neurophysiological methods, such as the nociceptive blink reflex (nBR) and visual evoked potentials (VEPs). These assessments provide information about the modulation of relevant stations in the trigemino-vascular system, specifically the trigemino-cervical complex and the occipital cortex.

Our study includes an evaluation of brain functional connectivity using High-Density Electroencephalography (HD-EEG). Recently, we analyzed potential variations in functional connectivity within the Resting State Network (RSN) in migraine patients undergoing six months of treatment with monoclonal antibodies targeting the CGRP pathway through serial HD-EEG evaluations (unpublished data). Our findings demonstrate that migraine patients, when compared to healthy controls, exhibit widespread hyperconnectivity in the theta and delta frequency bands, potentially attributable to dysfunction of the generators of these frequency bands, highlighting the importance of the thalamo-cortical dysrhythmia concept in migraine pathophysiology. Conversely, longitudinal comparisons revealed a trend towards normalization of connectivity in patients with a good clinical response to anti-CGRP monoclonal antibodies.

From a biochemical standpoint, our group has demonstrated that the gene expression of endocannabinoid catabolizing enzymes - fatty acid amide hydrolase (FAAH) and monoacylglycerol lipase (MAGL) - is altered in peripheral cells of patients with episodic and chronic migraine and is correlated with migraine severity. Similarly, various literature evidence supports the role of microRNAs in the mechanisms underlying migraines. Elevated expression levels of miR-382-5p and miR-34a-5p, combined with lower levels of miR-30a-5p expression, have been found in migraine patients compared to healthy controls, confirming an epigenetic alteration. In a previous study, we reported that peripheral levels of miR-382-5p and miR-34a-5p in migraine patients were correlated with disease severity, as they were increased in patients with chronic migraine and medication-overuse headache (CM-MOH) compared to episodic migraine (EM) patients, suggesting involvement in chronicization, while not excluding an influence of pharmacological migraine treatments . Elevated levels of miR-155, a microRNA known to modulate inflammation, have been found in peripheral cells of both EM and CM-MOH patients compared to healthy controls, with higher levels in chronic patients.

The overarching aim of this project is the identification of specific neurophysiological and biomolecular signatures that differentiate subjects with migraine who benefit or do not benefit from atogepant treatment. This aim will be achieved via a thorough neurophysiological and biochemical profiling of subjects with high frequency episodic migraine treated with atogepant 60 mg for a period of 3 months.

STUDY DESIGN:

Patients will be enrolled from those attending the outpatient clinic of IRCCS Mondino Institute (Pavia). The investigators will enroll 30 patients with high-frequency episodic migraine (8-14 monthly migraine days) with clinical indications to start atogepant (ATO - 60 mg daily) according to the Italian regulations.

The investigators will collect clinical data and perform biochemical and neurofunctional profiling of migraine patients at baseline (T0) and after three months of atogepant treatment (T1).

METHODS: All patients will undergo at T0 and T1:

1. Biochemical profiling that will include analysis of:

   * eCBome system: FAAH, MAGL mRNA in PBMCs;
   * plasma levels of CGRP, PACAP, and VIP;
   * miR-382-5p, miR-34a and miR-155 in PBMCs. The investigators will collect biochemical sampling between 9 and 11 a.m. to avoid circadian rhythm influence. All evaluation will be performed in the interictal phase.

   The following collection methods will be adopted: • mRNA and microRNA analysis in PBMCs. Blood samples will be collected within ethylenediamine tetra-acetic acid tubes, the investigators will first isolate PBMCs and total RNA. Ubiquitin C and U6 will act as housekeeping genes for genes coding for the eCBome enzymes and miRNAs. • CGRP alpha, PACAP-38 and VIP levels will be measured using a commercial enzyme linked immunosorbent assay.
2. Neurofunctional profiling that will include:

   * recording of the Nociceptive Withdrawal Reflex (RIII);
   * recording of the nociceptive Blink Reflex (nBR);
   * recording of High-Density EEG (HD-EEG);
   * recording of Visual Evoked Potentials (VEP). The following methods will be adopted: - Nociceptive Withdrawal Reflex (RIII reflex): The sural nerve will be stimulated via surface electrodes behind the right lateral malleolus. Reflex threshold (≥20 μV, >10 msec) will be determined using the ladder method. Temporal summation threshold (TST) will be assessed by increasing stimulus intensity (5 stimuli at 2 Hz) until facilitation of the reflex response appears. (De Icco et al., 2020).- Nociceptive Blink Reflex (nBR): nBR R2 response will be recorded using a concentric electrode above the supraorbital nerve and surface electrodes at the orbicularis oculi muscle. Habituation will be evaluated with 25 stimuli at varying frequencies, with area under the curve (AUC) calculated for 5 averaged blocks. Habituation index (HI) will reflect percentage change in AUC from the last to the first block. (Perrotta et al., 2017). - Visual Evoked Potentials (VEP) recording: VEP will be recorded during monocular stimulation using black-and-white checkered patterns. Components (N70, P100, N145) will be analyzed, and habituation will be defined as the percentage change in P100 amplitude between the last and first block. (Ambrosini et al., 2017). High Density Electroencephalography recording (HD-EEG): Recordings (128 channels, high-pass: 0.5 Hz, low-pass: 100 Hz) will include four 6-minute resting-state sessions (2 with eyes open, 2 with eyes closed). Frequency bands (delta to gamma) will be analyzed using a validated custom pipeline to reconstruct cortical/subcortical neural sources.

STATISTICAL ANALYSIS: Sample size calculation was performed for the primary outcome of ATOM project (namely compare the TST threshold of the RIII reflex between T0 and T1. From previous papers, preliminary data and experience of our research group, an expected difference between the means at T0 and T1 of 2 mA is inferred, with a standard deviation of 4 mA for both measurements. The comparison will be made by t test for paired data or corresponding nonparametric test (Wilcoxon Signed Rank Test), after performing a preliminary test on the normality of the data (Shapiro test). The investigators will consider a test power of β=0.8 and a 95% confidence. The suggested sample size is n=30. Regarding the co-primary outcome (Aim 2 - gene expression of MAGLs in PBMCs) a power analysis was performed, considering a significant difference between T0 and T1 of 5 RQ (standard deviation 4 and 10 respectively). Assuming a sample size of 30, the expected power is more than 80%.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 70;
* Diagnosis of episodic migraine according to ICHD-3 criteria;
* Monthly migraine days between 8 and 14 (high-frequency episodic migraine pattern) in the 3 months before screening;
* Individuals naïve to CGRP-targeted treatments;
* No more than one ongoing migraine preventive treatment with a stable dose for at least 3 months.

Exclusion Criteria:

* Contraindications to atogepant;
* History of serious psychiatric conditions;
* Diagnosis of other primary or secondary headaches (only sporadic tension-type headache is allowed);
* Medical conditions considered clinically significant by the investigator;
* Chronic pain conditions that need chronic treatment;
* Abuse of alcohol and/or drugs;
* Pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with high frequency episodic migraine attending the outpatient clinic of the Headache Science & Neurorehabilitation Center of the IRCCS Mondino Foundation (Pavia, Italy).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Temporal summation threshold of the RIII reflex (continuos variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Temporal summation threshold of the RIII reflex will be used to assess central sensitization after 3 months of treatment with atogepant 60 mg/day compared to baseline.
MAGL gene expression (continuos variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Changes in MAGL gene expression after 3 months of treatment with atogepant 60 mg/day

SECONDARY OUTCOMES:
Habituation index of the nociceptive Blink Reflex (continuous variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  "Habituation index" of the nociceptive Blink Reflex will be used to evaluate difference in brainstem habituation after three months of treatment with atogepant 60mg.
Habituation of the visual evoked potential (continuous variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Habituation of the visual evoked potential, assessed through P100 amplitude between the last and first block, will be used to assess changes in cortical habituation after three months of atogepant
Functional brain connectivity (continuous variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Changes in functional brain connectivity, assessed through HD-EEG after 3 months of treatment with atogepant 60 mg/day.
FAAH gene expression (continuous variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Changes in FAAH gene expression after 3 months of treatment with atogepant 60 mg/day.
Plasma levels of CGRP (continuous variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Changes in plasma levels of CGRP after 3 months of treatment with atogepant 60 mg/day.
Plasma levels of PACAP (continuous variable) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Changes in plasma levels of PACAP after 3 months of treatment with atogepant 60 mg/day.
Gene expression of miR-382-5p, miR-34a-5p, and miR-155 (continuous variables) | Baseline (T0) - three months of atogepant 60 mg treatment (T1)
  Changes in the gene expression of miR-382-5p, miR-34a-5p, and miR-155 after 3 months of treatment with atogepant 60 mg/day at the level of peripheral polymorphonuclear cells (PBMCs).

CONTACTS AND LOCATIONS:
Locations (1):
- Headache Science & Neurorehabilitation Center, Pavia, PAVIA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greco R, De Icco R, Demartini C, Zanaboni AM, Tumelero E, Sances G, Allena M, Tassorelli C. Plasma levels of CGRP and expression of specific microRNAs in blood cells of episodic and chronic migraine subjects: towards the identification of a panel of peripheral biomarkers of migraine? J Headache Pain. 2020 Oct 16;21(1):122. doi: 10.1186/s10194-020-01189-0. PMID 33066724
- [Background] Andersen HH, Duroux M, Gazerani P. Serum MicroRNA Signatures in Migraineurs During Attacks and in Pain-Free Periods. Mol Neurobiol. 2016 Apr;53(3):1494-1500. doi: 10.1007/s12035-015-9106-5. Epub 2015 Feb 1. PMID 25636687
- [Background] Greco R, Demartini C, Zanaboni AM, Tumelero E, Icco R, Sances G, Allena M, Tassorelli C. Peripheral changes of endocannabinoid system components in episodic and chronic migraine patients: A pilot study. Cephalalgia. 2021 Feb;41(2):185-196. doi: 10.1177/0333102420949201. Epub 2020 Sep 23. PMID 32967434
- [Background] Greco R, Demartini C, Zanaboni AM, Francavilla M, De Icco R, Ahmad L, Tassorelli C. The endocannabinoid system and related lipids as potential targets for the treatment of migraine-related pain. Headache. 2022 Mar;62(3):227-240. doi: 10.1111/head.14267. Epub 2022 Feb 18. PMID 35179780
- [Background] de Tommaso M, Ambrosini A, Brighina F, Coppola G, Perrotta A, Pierelli F, Sandrini G, Valeriani M, Marinazzo D, Stramaglia S, Schoenen J. Altered processing of sensory stimuli in patients with migraine. Nat Rev Neurol. 2014 Mar;10(3):144-55. doi: 10.1038/nrneurol.2014.14. Epub 2014 Feb 18. PMID 24535465
- [Background] Ambrosini A, Kisialiou A, Schoenen J. Visual and auditory cortical evoked potentials in interictal episodic migraine: An audit on 624 patients from three centres. Response to the letter by Omland et al. Cephalalgia. 2017 Oct;37(12):1209-1210. doi: 10.1177/0333102416680616. Epub 2016 Nov 21. No abstract available. PMID 27872339
- [Background] Perrotta A, Anastasio MG, De Icco R, Coppola G, Ambrosini A, Serrao M, Sandrini G, Pierelli F. Frequency-Dependent Habituation Deficit of the Nociceptive Blink Reflex in Aura With Migraine Headache. Can Migraine Aura Modulate Trigeminal Excitability? Headache. 2017 Jun;57(6):887-898. doi: 10.1111/head.13111. Epub 2017 May 10. PMID 28488755
- [Background] Coppola G, Di Lorenzo C, Schoenen J, Pierelli F. Habituation and sensitization in primary headaches. J Headache Pain. 2013 Jul 30;14(1):65. doi: 10.1186/1129-2377-14-65. PMID 23899115
- [Background] De Icco R, Fiamingo G, Greco R, Bottiroli S, Demartini C, Zanaboni AM, Allena M, Guaschino E, Martinelli D, Putorti A, Grillo V, Sances G, Tassorelli C. Neurophysiological and biomolecular effects of erenumab in chronic migraine: An open label study. Cephalalgia. 2020 Oct;40(12):1336-1345. doi: 10.1177/0333102420942230. Epub 2020 Jul 26. PMID 32715736
- [Background] De Icco R, Greco R, Demartini C, Vergobbi P, Zanaboni A, Tumelero E, Reggiani A, Realini N, Sances G, Grillo V, Allena M, Tassorelli C. Spinal nociceptive sensitization and plasma palmitoylethanolamide levels during experimentally induced migraine attacks. Pain. 2021 Sep 1;162(9):2376-2385. doi: 10.1097/j.pain.0000000000002223. PMID 33587406
- [Background] Lipton RB, Pozo-Rosich P, Blumenfeld AM, Li Y, Severt L, Stokes JT, Creutz L, Gandhi P, Dodick D. Effect of Atogepant for Preventive Migraine Treatment on Patient-Reported Outcomes in the Randomized, Double-blind, Phase 3 ADVANCE Trial. Neurology. 2023 Feb 21;100(8):e764-e777. doi: 10.1212/WNL.0000000000201568. Epub 2022 Nov 17. PMID 36396451
- [Background] Rissardo JP, Caprara ALF. Gepants for Acute and Preventive Migraine Treatment: A Narrative Review. Brain Sci. 2022 Nov 24;12(12):1612. doi: 10.3390/brainsci12121612. PMID 36552072
- [Background] Pozo-Rosich P, Ailani J, Ashina M, Goadsby PJ, Lipton RB, Reuter U, Guo H, Schwefel B, Lu K, Boinpally R, Miceli R, De Abreu Ferreira R, McCusker E, Yu SY, Severt L, Finnegan M, Trugman JM. Atogepant for the preventive treatment of chronic migraine (PROGRESS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Sep 2;402(10404):775-785. doi: 10.1016/S0140-6736(23)01049-8. Epub 2023 Jul 26. PMID 37516125
- [Background] Goadsby PJ, Dodick DW, Ailani J, Trugman JM, Finnegan M, Lu K, Szegedi A. Safety, tolerability, and efficacy of orally administered atogepant for the prevention of episodic migraine in adults: a double-blind, randomised phase 2b/3 trial. Lancet Neurol. 2020 Sep;19(9):727-737. doi: 10.1016/S1474-4422(20)30234-9. PMID 32822633
- [Background] Ailani J, Lipton RB, Goadsby PJ, Guo H, Miceli R, Severt L, Finnegan M, Trugman JM; ADVANCE Study Group. Atogepant for the Preventive Treatment of Migraine. N Engl J Med. 2021 Aug 19;385(8):695-706. doi: 10.1056/NEJMoa2035908. PMID 34407343
- [Background] Buse DC, Armand CE, Charleston L 4th, Reed ML, Fanning KM, Adams AM, Lipton RB. Barriers to care in episodic and chronic migraine: Results from the Chronic Migraine Epidemiology and Outcomes Study. Headache. 2021 Apr;61(4):628-641. doi: 10.1111/head.14103. Epub 2021 Apr 1. PMID 33797078